CLINICAL TRIAL: NCT06770933
Title: A Phase II, Double-Masked, Randomised, Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety of Orally Administered VX-01 in Diabetic Retinopathy OF Non-Proliferative Type (NPDR)
Brief Title: A Study to Evaluate the Efficacy and Safety of Orally Administered VX-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vantage Biosciences Ltd (Industry)
Collaborators: Vantage Biosciences Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX01-DR-201
Record Dates: First submitted 2024-12-16; First posted 2025-01-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy; NPDR - Non Proliferative Diabetic Retinopathy
Keywords: NPDR; Diabetic Retinopathy; AOC3; VAP-1; SSAO; VAP1; Amine Oxidase Copper containing 3; Amine Oxidase; HPAO
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: This is a multi-center, double-masked, randomized, placebo-controlled, parallel group study, where subjects will be randomized 1:1 to 1 of 2 study cohort of VX-01 and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- VX-01 (Experimental): Cohort 1 will include 50 subjects who will be randomized to take investigational drug VX-01 (film-coated tablets) at dose of 150 mg, administered BID.
  Interventions: Drug: VX-01
- Placebo (Placebo Comparator): Cohort 2 will include 50 subjects who will be randomized to receive the placebo drug (film-coated tablets), that will be administered BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-01 — There is no physical difference in VX-01 and the placebo. The only difference lies in active ingredient found in VX-01, which is the compound that will be evaluated in the course of this study.
  Arms: VX-01
Drug: Placebo — Placebo will be supplied as a tablet identical to test drug but without VX-01. Placebo packaging will be identical to IP in order to keep study personnel and subjects masked.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of VX-01 as stand-alone treatment for Diabetic Retinopathy of Non-Proliferative Type (NPDR).

The primary objective of the study is to evaluate the efficacy of daily oral doses of VX-01 versus placebo following 52 weeks of treatment.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, double-masked, randomized, placebo-controlled, parallel group study to evaluate the efficacy of oral doses of VX-01 in subjects with moderate to severe NPDR, without CI-DME.

Approximately 100 male and female subjects aged ≥ 18 years with a documented diagnosis of Type 1 Diabetic Mellitus or Type 2 Diabetic Mellitus with moderate to severe NPDR (without CI-DME) will be enrolled, if they meet all the eligibility criteria for the study.

Subjects will be randomized 1:1 to 1 of 2 study cohorts:

* Cohort 1 (n = 50): VX-01 (film-coated tablets, 150 mg administered BID)
* Cohort 2 (n = 50): Placebo (film-coated tablets, administered BID)

Subjects will be stratified by the presence or absence of proliferative diabetic retinopathy (PDR) and by glycated hemoglobin (HbA1c) of ≥ 8.5% or < 8.5% at Screening. All subjects will take 1 tablet of VX-01 or placebo BID for 52 consecutive weeks. All subjects will be followed for 12 weeks after completion of treatment at Week 52.

The Sponsor, study site staff, monitors, personnel, and subjects will be masked to treatment assignment during the entirety of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject prior to any study-related procedures.
* Subject must be aged > 18 years at the time of Screening.
* Subject must have a body mass index (BMI) of between 18 and 40 kg/m2, inclusive.
* Subject has a documented diagnosis of T1DM or T2DM.
* Subject has moderate to severe NPDR, as determined by a Central Reading Centre (CRC) using DRSS in at least one eye
* Subject must have clear ocular media and be able to undergo adequate pupil dilation to allow adequate fundus imaging of both eyes.
* Female subject must be either:

  1. Of non-childbearing potential: post-menopausal or documented surgically sterile post hysterectomy (at least 1 month prior to Screening)
  2. Or, if of childbearing potential, must have a negative serum pregnancy test at Screening and must use 2 acceptable forms of contraception, starting at Screening and throughout the study period and for 28 days after the final IP administration.
* Female subject must not be breastfeeding at Screening or during the study period, and for 28 days after the final IP administration.
* Male subject must be surgically sterile (> 30 days since vasectomy with no viable sperm), or if engaged in sexual relations with a female of childbearing potential, the couple should agree to use 2 acceptable contraceptive methods from Screening, during the study, and for 28 days after last IP administration.

Female subject must not donate ova or male subject must not donate sperm starting at Screening and throughout the study period, and for 28 days after the final IP administration.

* Subject must have Best Corrected Visual Acuity (BCVA) assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) protocol letters score of ≥ 70 letters in study eye, and ≥ 20 letters in the non-qualified fellow eye.
* Subject must have the ability, in the opinion of the Investigator, and willingness to return for all scheduled visits and perform all assessments.
* Subject agrees not to participate in another interventional study after signing the informed consent and until the End of Study (EOS) visit has been completed.

Exclusion Criteria:

Ophthalmic:

* Presence of CI-DME (with central subfield thickness [CST] measured greater than 325 μm on spectral domain optical coherence tomography [SD-OCT]) threatening the center of the macula (within 1,000 μm of the foveal center) in either eye, or presence of DME requiring treatment.
* Presence of moderate to high-risk PDR (DRSS level 65 or higher).
* Any prior treatment (in either eye) with:

  1. Focal or grid laser photocoagulation within the past 6 months prior to Screening or pan-retinal photocoagulation (PRP) at any time.
  2. Systemic or intravitreal anti-vascular endothelial growth factor (VEGF) agents within the last 12 months prior to Screening.
  3. Intraocular, sub-tenon or periocular steroids, including triamcinolone and dexamethasone implant within the last 6 months, or suprachoroidal triamcinolone within the last 3 months prior to Screening.
  4. Fluocinolone implant within the last 3 years prior to Screening.
  5. Prior treatment for NPDR with any other treatment which is not labelled for NPDR within 1 year prior to Screening (e.g., calcium dobesilate, fibrate medication).
  6. Vitrectomy at any timepoint prior to Screening.
  7. Yttrium-Aluminium-Granate (YAG) capsulotomy within 3 months prior to Screening.
* Active uveitis, vitritis, or infection in either eye including infectious conjunctivitis, keratitis, scleritis, or endophthalmitis.
* History of corneal transplant and/or vitrectomy or any other ocular incisional surgery in either eye (e.g., shunt surgery). Note: Subjects who have had cataract or refractive surgery in either that was more than 3 months prior to Screening may be permitted at the discretion of the Investigator.
* Uncontrolled glaucoma, as evidenced by intraocular pressure (IOP) > 25 mmHg despite up to 4 glaucoma medications, or evidence of glaucomatous visual field loss or has advanced glaucoma (e.g., prior shunt surgery) in either eye.
* Clinically significant ocular disease in either eye that in the opinion of the Investigator would preclude participation in the study.
* Presence of macular or retinal vascular disease including DME and/or retinopathy from causes other than diabetes, age-related macular degeneration, pattern dystrophy, choroidal neovascularisation of any cause, retinal vein occlusion, retinal artery occlusion in either eye.
* History of retinal detachment or full-thickness macular hole post intraocular surgery in either eye, or idiopathic or autoimmune uveitis in either eye.
* Any other ocular disease that may cause substantial reduction in BCVA.

Systemic:

* Known, suspected hypersensitivity or contraindication to IP.
* Uncontrolled diabetes mellitus with HbA1c of ≥ 12%.
* Initiation of treatment with glucagon-like peptide-1 (GLP-1) modulators for glycaemic control and other indications within the last 3 months prior to Screening.
* Initiation of intensive insulin treatment (a pump or multiple daily injections) within 3 months prior to Screening or plans to do so in the next 3 months.
* Current use of coumarin anticoagulants (Coumadin/Warfarin).
* On dialysis or an estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73m2 as per CKD-EPI evaluation at Screening. (Active Diabetic Ketoacidosis or Hyperglycemic Hyperosmolar Nonketotic State).
* Hypertension with resting diastolic blood pressure (BP) > 100 mmHg or systolic BP > 180 mmHg on 2 consecutive measurements at least 5 minutes apart. Note: If the result is out of range, the assessment may be repeated once prior to randomisation for confirmation.
* Resting heart rate outside the specified range (50 to 110 beats per minute). Note: If the result is out of range, the assessment may be repeated once prior to randomisation for confirmation.
* History of chronic liver disease or presence of elevated (defined as > 3 × upper limit of normal) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) consistent with such diagnosis.
* Known to be immunocompromised or receiving immunosuppressive therapy. Note: Subjects receiving low dose corticosteroids may be eligible, at the discretion of the Investigator.
* Currently receiving treatment with a strong inhibitor of the P-glycoprotein transporter (see Section 6.4.2), which may interfere with the IP.
* History of allergy to fluorescein.
* Any disease or medical condition that in the opinion of the Investigator would interfere with the study, prevent the subject from successfully participating in the study, or which might confound the study results.
* Participation in any investigational study within 30 days prior to Screening or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion.
* History of blood transfusion or severe blood loss within 3 months prior to Screening, known hemoglobinopathy, and severe anaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of oral doses of VX-01 in subjects compared to placebo following 1 year of treatment. | From enrollment to the end of treatment at week 52
  The endpoint of this objective is the proportion of subjects who do not develop a worsening from Baseline in binocular ETDRS DRSS at Week 52. The diabetic retinopathy severity scale (DRSS) is a scale healthcare professionals use to measure the severity and progression of a person's diabetic retinopathy. The main DRSS is the Early Treatment Diabetic Retinopathy Study (ETDRS) scale which will be used in this study.

SECONDARY OUTCOMES:
To evaluate the efficacy of VX-01 in subjects with moderate to severe NPDR without CI-DME by determining the overall change from Baseline in BCVA letter scores. | From enrollment to the end of treatment at week 52
  Endpoint measurement of this objective will be improvement in Best Corrected Visual Acuity (BCVA), i.e. higher scoring at end of treatment compared to enrollment (baseline).
To evaluate the efficacy of VX-01 in subjects with moderate to severe NPDR without CI-DME by determining the overall change from Baseline in the ETDRS DRSS scores. | From enrollment to the end of treatment at week 52
  Endpoint measurement of this objective will be improvement in the Early Treatment Diabetic Retinopathy score (ETDRS), i.e. higher score at end of treatment compared to enrollment (baseline measure)
Incidence of Treatment-Emergent Adverse Events (TEAEs) when taking multiple oral doses of VX-01. | From enrollment to the end of treatment at week 52
  Endpoint measurement of this objective will include assessing the nature, frequency, and severity of systemic and ocular TEAEs across the duration of the study. A lower number of TEAEs would point towards a better safety and tolerability profile of VX-01
Number of subjects developing moderate to high risk proliferative diabetic retinopathy | From enrollment to the end of treatment at week 52
  Measurement of proportion of subjects who develop moderate to high-risk proliferative diabetic retinopathy in either eye at Week 24 and also at Week 52 will be quantified. This will aid in understanding the safety of VX-01.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (8):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - California Retina Consultants- Santa Barbara, Santa Barbara, California
  - Florida Retina Institute - Jacksonville Southside, Jacksonville, Florida
  - Retina Associates, Elmhurst, Illinois
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Erie Retina Research, Erie, Pennsylvania
  - Piedmont Eye Center, Lynchburg, Virginia
- Australia (8):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - Retina And Eye Consultants Hurstville, Hurstville, New South Wales
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - University of the Sunshine Coast Clinical Trials (Birtinya), Birtinya, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Hong Kong (2):
  - Prince of Wales Hospital The Chinese University of Hong Kong, Shatin
  - HKU Eye Centre, Wong Chuk Hang
- Malaysia (5):
  - University Malaya Medical Centre, Petaling Jaya, Kuala Lumpur Federal Territory of Kuala Lumpur
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Shah Alam, Shah Alam, Selangor
  - Hospital Al-sultan Abdullah Uitm, Sungai Buloh, Selangor
  - Hospital Selayang, Selayang Baru Utara
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided